CLINICAL TRIAL: NCT00535054
Title: An Open Study to Assess the Safety and Patients' Satisfaction Tears Again* in the Treatment of Dry Eye Symptoms
Brief Title: Study to Assess the Safety and Patients' Satisfaction of Tears Again* in the Treatment of Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trima, Israel Pharmaceutical Products (Industry)
Responsible Party: David Zadok, MD, Department of Ophthalmology, Assaf Harofeh Medical Center,Zerifin, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06.11
Record Dates: First submitted 2007-09-23; First posted 2007-09-26 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tears Again (Experimental): All subjects shall be treated with Tears Again.
  Interventions: Drug: Tears Again

INTERVENTIONS:
Drug: Tears Again — Liposome Eye Spray

SUMMARY:
The purpose of this study is to determine safety and patients' satisfaction when using Tears Again to treat Dry Eye Symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Suffer from at least two of the following ocular symptoms: burning, stinging, excessive tearing, dryness, grittiness, foreign body sensation ( including patients suffering from blepharitis).
* Use artificial tears or any other treatment for these symptoms three or more times a day.

Exclusion Criteria:

* Known hypersensitivity to Phenoxyethanol.
* Pregnant and lactating women.
* Receive other ophthalmic medication (except for eyelid hygiene preparations).
* Graft-versus-host disease patients.
* Participated during the last month in another clinical trial.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Schirmer Test, Lissamine Green Test and BUT. | On enrollment and one month later.

SECONDARY OUTCOMES:
Questionaire | One, three and four weeks after treatment commencement.

CONTACTS AND LOCATIONS:
Overall Officials: David Zadok, MD, Principal Investigator — Department of Ophthalmology, Assaf Harofeh Medical Center,
Locations (1):
- Department of Ophthalmology, Assaf Harofeh Medical Center,, Ẕerifin, Israel

REFERENCES:
- [Background] Lee S, Dausch S, Maierhofer G, Dausch D. [A new therapy concept for the treatment of dry eye--the usefulness of phospholipid liposomes]. Klin Monbl Augenheilkd. 2004 Oct;221(10):825-36. doi: 10.1055/s-2004-813715. German. PMID 15499517
- [Background] Dausch D, Lee S, Dausch S, Kim JC, Schwert G, Michelson W. [Comparative study of treatment of the dry eye syndrome due to disturbances of the tear film lipid layer with lipid-containing tear substitutes]. Klin Monbl Augenheilkd. 2006 Dec;223(12):974-83. doi: 10.1055/s-2006-927266. German. PMID 17199193